CLINICAL TRIAL: NCT06808997
Title: Criteria and Reasons for Extubation and Non-extubation in Preterm Infants: A Mixed Methods Study Prospectively Exploring Extubation and Reintubation Practices in Extremely Preterm Infants, and Associated Respiratory Outcomes.
Brief Title: Prospective Multicentre Mixed Methods Study to Explore Extubation Practices and Respiratory Outcomes in Extremely Preterm Neonates.
Acronym: CERAINE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: CERAINE
Record Dates: First submitted 2025-01-13; First posted 2025-02-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: PreTerm Neonate; Extubation Readiness; Extubation Failure; Respiratory Morbidity; Bronchopulmonary Dysplasia; Mechanical Ventilation
Keywords: extremely preterm infants; extubation; mechanical ventilation; bronchopulmonary dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extremely Low Gestational Age Newborns (elgans): No intervention. unique group.

SUMMARY:
The purpose of this observational study is to learn about neonatologists' perceptions of extubation readiness and extubation and reintubation practices in extremely preterm infants in the first 2 weeks of life using prospective qualitative and quantitative data. Actual extubation readiness is defined as successful extubation, defined as no reintubation in the 7 days following extubation.

Key research questions are: How do clinicians assess extubation readiness in this population? Does this assessment correlate with actual extubation success? What factors (reasons, clinical status, ventilatory parameters) are associated with extubation readiness? Patients born before 28 weeks gestational age and admitted to the neonatal intensive care unit (NICU) within the first 24 hours are be included. The attending physician will complete a prospectively administered questionnaire with open-ended and multiple-choice questions to daily assess the decision and rationale for extubation or non-extubation of patients mechanically ventilated during the first 15 days of life.

Patient characteristics, respiratory outcomes, and mortality will be recorded until the end of hospitalisation and/or definitive weaning from any ventilatory support or supplemental oxygen.

DETAILED DESCRIPTION:
With prolonged stays in the neonatal intensive care unit (NICU) and significant respiratory morbidity, respiratory management of the most premature newborns - born before 28 weeks gestational age (GA) - brings a number of challenges. Despite recommendations to give priority to non-invasive ventilation in cases of respiratory insufficiency, recent studies show that over 80% of these newborns receive mechanical ventilation (MV) at least once in their NICU course, most within the first week of life (100% if born at 23 SA, >90% at 24 and 25 SA, >80% at 26 and >70% at 27 weeks GA). Several studies have shown that a longer cumulative duration of MV is associated with a worse respiratory and neurodevelopmental prognosis in this population.

Early extubation is therefore recommended. However, extubation failures in patients born at these early stages of life are common and are per se associated with respiratory morbidity. Extubation failure is defined in the literature as reintubation within days of extubation.

A delay of 7 days after extubation has been identified as the time frame for capturing extubations related to respiratory causes. In a French study, using the SEPREVEN cohort for patients born before 27 weeks' GA, extubation failure at 3, 7 and 15 days concerned 25%, 33% and 50% of patients respectively. The decision to extubate a premature patient is a complex one, but contributes in part to the patient's outcome.

Shalish referred to the concept of "extubation readiness dilemma" to indicate the uncertainty surrounding the clinical features associated with successful extubation. Identifying a state for each patient that allows successful extubation, without reintubation in the following days, is most often based on ward routines in which assessments of the infant's respiratory capacity are taken into account. Medical literature doesn't provide recommendations on extubation criteria, and practices differ from one unit to another.

The aim of this study is to provide a detailed description of extubation practices and failures in several NICUs in France, based on a prospective collection of qualitative and mixed data.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 28 weeks of gestation
* Age at admission to the participating unit <24 hours

Exclusion Criteria:

* Parental opposition to their infant's clinical data collection
* Participation in a research protocol with potential impact on extubation and/or duration of mechanical ventilation

Ages: 1 Minute to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participation in the study is proposed to type 3 neonatal intensive care units in France. Extremely premature newborns born before 28 weeks gestation in the participating units will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Reasons for non-extubation in case of MV in patients born before 28 wks GA in the first 15 days of life, | On a 12 hours basis from Day 0 to Day 2 of life, and on a dialy basis from Day 2 to Day 15 of life (according to the period the patient is on Mechanical Ventilation)
  For each included patient who is intubated and mechanically ventilated during a period within his first 15 days of life, the reasons for non-extubation. These are the reasons reported by the physician by answering a qualitative questionnaire with an open-ended question, and preexistent possible multiple choices.

SECONDARY OUTCOMES:
Reported perceived extubation readiness in Extremely Low Gestational Age Neonates (ELGANs) born before 28weeks gestation and mechanically ventilated in a period within the first 15 days of life. | These data will be collected in case of Mechanical Ventilation every 48 hours between the Birthday and Day 2 of life and then every morning between Day 2 and Day 15 of life
  Reported perceived extubation readiness in ELGANs born before 28weeks gestation and mechanically ventilated in a period within the first 15 days of life, defined as Reasons for extubation and ventilatory and clinical data,
Occurrence of Extubation failure in ELGANs on Mechanical ventilation within the first 15 days of life. | These data will be collected in case of Mechanical Ventilation every 48 hours between the Birthday and Day 2 of life and then every morning between Day 2 and Day 15 of life
  Occurrence of Extubation failure defined as reintubation in the 7 days after an extubation.
Corrected gestational age on definitive discontinuation of MV, of Positive Pressure Non-Invasive Ventilation (NIV), of High Flow Nasal Cannula (HFNC) ventilation) and Low Flow Nasal Cannula Ventilation (LFNNC) | From the day of birth to 4 months of age.
  Corrected gestational age on definitive discontinuation of MV, of Positive Pressure Non-Invasive Ventilation (NIV), of High Flow Nasal Cannula (HFNC) ventilation) and Low Flow Nasal Cannula Ventilation (LFNNC)
Cumulative duration of mechanical ventilation (MV) during the NICU stay. | These data will be collected from the day of birth to the day of discharge from the NICU, up to maximum 4 months of age..
  Sum of the days of mechanical ventilation during the NICU stay, collected prospectively.
The cumulative duration of any respiratory support | From the day of birth to the day of discharge from the hospital, up to maximum 4 months of age.
  The cumulative duration of positive pressure Non-Invasive Ventilation (PPNIV) and High Flow Nasal Ventilation (HFNV), Low Flow Nasal Ventilation (LFNV) during the entire hospital stay
Duration of Mechanical Ventilation and Positive Pressure Non-Invasive Ventilation | From the day of birth to the day of discharge from the hospital, up to 4 months of age
  Sum of the days of Mechanical Ventilation or positive pressure non invasive ventilation during the entire hospital stay
Bronchopulmonary dysplasia at 36 weeks corrected Gestational Age | At 36 weeks corrected gestational age
  Bronchopulmonary dysplasia at 36 weeks corrected Gestational age defined as need for any type of ventilation (invasive or non-invasive) or low flow oxygen therapy at 36 weeks gestational age.
Mortality | From the day of birth to the day of discharge from the hospital, maximum 5 months of age
  Mortality before discharge from the hospital
Length of stay in the Neonatal Intensive Care Unit (NICU) | From the day of birth to the day of discharge from the NICU, maximum 4 months of life
  Length of stay in the NICU
Factors involved in the perception of "too altered respiratory condition to be extubated" | From the day of birth to day 15 of life during the period on Mechanical Ventilation
  Description of the reasons related to the respiratory system, clinical respiratory conditions (e;g. apneas ....) and ventilatory settings (pressure, oxygen, ...) reported by the physician associated with a reported "too altered respiratory condition to be extubated" condition.
Clinician-reported Prognosis of extubation succes | From day of birth to day 15 of life during the period on Mechanical Ventilation
  Physician-reported prognosis of extubation based on a 4 points scale (from 1 "unconfident" to 4 "very confident")
Description of complications of intubation | from the day birth to the day discharge from the NICU, up to maximum 4 months of life
  Description of a multiple choice of complications after each intubation :
  No complication, oropharyngeal lesion, cardiorespiratory arrest, severe intraventricular haemorraghe, contribution to patient's death.

OTHER OUTCOMES:
Description of unit practices (mechanical ventilation weaning protocol and/or extubation criteria in standard care) | From the date of enrollment to the date of the end of the inclusions, which means one year.
  Description of unit practices (use of a Mechanical Ventilation weaning protocol and/or the use of extubation criteria in standard care)

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - Dr Jean-michel Roue, Brest, Brest
  - CHU Amiens Sud, Amiens
  - CH Cote Basque, Bayonne
  - CHU De Besancon, Besançon
  - Hopital Femme Mére Enfant - HFME, Bron
  - Centre Hospitalier Public du Cotentin, Cherbourg-Octeville
  - CH Estaing, Clermont-Ferrand
  - Chu Louis Mourier, Colombes
  - CHIC, Créteil
  - CHU Grenoble Alpes _site nord, Grenoble
  - CHU Félix Guyon, La Réunion
  - CHU Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHU Lille, Lille
  - HME Limoges, Limoges
  - APHM_ Hôpital Nord, Marseille
  - GHEF- Site de MEAUX, Meaux
  - Chi Andre Gregoire, Montreuil
  - GHRMSA-Hopital Emile Muller, Mulhouse
  - CHU NICE, Nice
  - Chu Nimes, Nîmes
  - CH Orléans, Orléans
  - CHU Robert Debre, Paris
  - Chu Port Royal, Paris
  - CHU Necker, Paris
  - CHI Poissy - St Germain en LayE, Poissy
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CH General Delafontaine, Saint-Denis
  - CH GHPSO, Senlis
  - CH Troyes, Troyes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shalish W, Keszler M, Davis PG, Sant'Anna GM. Decision to extubate extremely preterm infants: art, science or gamble? Arch Dis Child Fetal Neonatal Ed. 2022 Jan;107(1):105-112. doi: 10.1136/archdischild-2020-321282. Epub 2021 Feb 24. PMID 33627331